CLINICAL TRIAL: NCT06498362
Title: The "New" Place of LEVETIRACETAM in the Management of Status Epilepticus in Children: Multicenter Retrospective Study on 151 Children Over Three Months Old
Brief Title: The "New" Place of LEVETIRACETAM in the Management of Status Epilepticus in Children
Acronym: LEVET
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9067
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy in Children
Keywords: Epilepsy; Epilepsy in Children
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Status epilepticus is the leading neurological emergency in children, with mortality 2-7% and significant morbidity (10-20%). It is defined as the occurrence of a crisis lasting more than 5 minutes and requiring the implementation of treatment to stop it and thus limit the immediate and long-term consequences.

The research hypothesis is that LEVETIRACETAM is non-inferior to PHENYTOIN in terms of cessation and absence of recurrence of status epilepticus, with better clinical tolerance in children from 3 months to 17 years old, with or without epileptic disease, with or without a history of status epilepticus

ELIGIBILITY:
Inclusion Criteria:

* Minor patient aged 3 months to 17 years
* 2nd line treatment with LEVETIRACETAM or PHENYTOIN after failure of benzodiazepines
* Supported in one of the participating centers during the period from November 1, 2019 to May 31, 2023
* Subject or parents who have not expressed, after information, their opposition to the reuse of their data for the purposes of this research.

Exclusion Criteria:

* Patient or parents having expressed their opposition to participating in the study.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor patient aged 3 months to 17 years having 2nd line treatment with LEVETIRACETAM or PHENYTOIN after failure of benzodiazepines
Sampling Method: Non-Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Highlight non-inferiority of LEVETIRACETAM compared to PHENYTOIN | Up to 2 years
  The non-inferiority of LEVETIRCETAM in comparison with PHENYTOIN is based on a composite primary endpoint consisting of the total duration of the seizure, the need for another antiepileptic treatment to resolve the seizure or recurrence within 24 hours. following the start of treatment for a new status epilepticus and the total duration of hospitalization.
  The need for another antiepileptic drug or recurrence is a binary variable with presence (= yes = 1) or absence (= no = 0).
  The total duration of the crisis is expressed in minutes, and corresponds to the interval between the identification of the event and the objectification of its cessation.
  The total duration of hospitalization is expressed in days, and corresponds to the duration between the first day of hospitalization (regardless of the location) and the day of discharge (regardless of the department).

CONTACTS AND LOCATIONS:
Locations (1):
- Service pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France